CLINICAL TRIAL: NCT00686270
Title: A Phase 3, Open Label 96-week Extension Study of the Safety of Apricitabine in Treatment-experienced HIV-1 Infected Patients Who Have Completed Protocol AVX-301 or AVX-302 or Who Have Met the Criteria for Open-label Access to ATC Because of Virological Failure/Lack of Response
Brief Title: A Long Term Safety Study of Apricitabine in HIV-infected Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was withdrawn owing to Sponsor decision
Sponsor: Avexa (Industry)
Responsible Party: Susan Cox, Avexa Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVX-303
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; NRTI resistance; M184V mutation; reverse transcriptase; apricitabine; drug resistance; safety and tolerability; therapy failure; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — apricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): apricitabine
  Interventions: Drug: apricitabine

INTERVENTIONS:
Drug: apricitabine — Initially 1200mg apricitabine twice daily orally. Following the determination of the optimum dose (800mg or 1200mg twice daily) in the pre-ceeding study AVX-301,patients may be switched to the optimum dose,if required.
  Other Names: ATC; AVX754

SUMMARY:
This study will examine the long term safety of apricitabine in HIV-1 infected patients from studies AVX-301 or AVX-302. Eligible patients are those who have either (a)completed studies AVX-301 or AVX-302; or (b)met the criteria for virological failure/lack of response, and consequently wish to withdraw early from studies AVX-301 or AVX-302.

DETAILED DESCRIPTION:
The clinical study AVX-301 studies the efficacy and safety of 800mg and 1200mg BID ATC in combination with an optimized background in patients who are HIV-1 infected and have failed treatment with emtricitabine or lamivudine and have confirmed M184V/I mutation. Patients who do not achieve at least a 0.5 log10 copies/mL decrease in plasma HIV RNA by Week 16, or who experience a >1.0 log10 copies/mL increase (confirmed on two separate occasions at least one week apart) in plasma HIV RNA from nadir at or after Week 16, are eligible for screening for entry into this study. In addition, patients who complete study AVX-301 are also eligible for screening. The clinical study AVX-302 is similar and studies the efficacy and safety of a single dose of ATC (determined in AVX-301). Patients in AVX-302 who experience virologic failure or lack of virologic response will similarly be eligible for screening for entry into this study. In addition, patients who complete study AVX-302 are also eligible for screening. This is a phase 3, open-label, multi-center study of up to 96 weeks duration. Patients will receive for up to 96 weeks open-label ATC, initially at a dose of 1200mg orally BID. Following selection of the optimum ATC dose in protocol AVX-301 and termination of one of the two ATC doses (800mg or 1200mg orally BID) in protocol AVX-301, patients in this protocol will be transferred to the optimum dose, if required. The total number of patients expected to be enrolled in studies AVX-301 and AVX-302 is approximately 1866 in total.Patients will receive ATC orally in combination with their existing ART. Background antiretroviral therapy (ART) may be revised at any time during the study at the discretion of the investigator but must not include lamivudine, emtricitabine, zalcitabine or any other deoxycytidine analogue NRTI. The study will examine the safety and tolerability of long term treatment with apricitabine in combination with other ART.

ELIGIBILITY:
Inclusion Criteria:

* Patients who complete studies AVX-301 or AVX-302 or :Patients who meet the criteria for virologic failure/lack of response in study AVX-301 or AVX-302
* 18 years of age, or older
* Male, or non-pregnant, non-breastfeeding female patients, who agree to comply with the applicable contraceptive requirements of the protocol.

Exclusion Criteria:

* Prior withdrawal from AVX-301 or AVX-302
* Current acute or chronic hepatitis B virus infection
* Current treatment for hepatitis C virus infection
* Renal Function not adequate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The number, type and severity of SAEs occuring during the study | Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Mike Saag, Professor, Principal Investigator — UAB Centre for AIDS Research, Birmingham, Alabama, 35294-2050, USA; Susan W Cox, PhD, Study Director — Avexa Ltd